CLINICAL TRIAL: NCT04139083
Title: The Clinical and Urodynamic Effects of Transvaginal or Laparoscopic Mesh Suspension for the Treatment of Pelvic Organ Prolapse
Brief Title: The Clinical Outcome of TVM or LSC Mesh Suspension for POP
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20190015
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Transvaginal mesh; Laparoscopic mesh suspension
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TVM group: Women with mainly uterine prolapse stage II or greater as defined by the POP-Q staging system treated with TVM
  Interventions: Procedure: TVM
- LSC mesh suspension group: Women with mainly uterine prolapse stage II or greater as defined by the POP-Q staging system treated with LSC mesh suspension
  Interventions: Procedure: LSC mesh suspension

INTERVENTIONS:
Procedure: LSC mesh suspension — Long mesh, a synthetic T-shaped mesh (Gynemsh, Ethicon, San Lorenzo, Puerto Rico), is delivered into the pelvic cavity. Bilateral mesh arms are extracted outside trocar wounds bilaterally to stabilize mesh position. The center piece is fixed to the cervix with 5mm ProTack screws (Covidien, New Haven, Connecticut). Fixation is strengthened with Stratafix 2-0 sutures (Ethicon, Norderstedt, Germany), followed by Tisseel fibrin sealant (Baxter, Deerfield, Illinois) for better hemostasis among surrounding tissues. An extraperitoneal tunnel is created along the left round ligament until reaching 2cm medial to the anterior superior iliac spine (ASIS). One arm of the long mesh is pulled out along the tunnel underneath round ligament and fixed with the fascia of oblique abdominis. The same procedure is repeated for the contralateral side. Bilateral round ligaments and the mesh arms are sutured continuously with Stratafix 2-0.
  Groups: LSC mesh suspension group
Procedure: TVM — Transvaginal mesh kit is delivered into the pelvis via vagina route.
  Groups: TVM group

SUMMARY:
The investigators aim to assess the surgical outcomes of transvaginal mesh (TVM) and laparoscopic (LSC) mesh suspension. During the study period, all women with main uterine prolapse stage II or greater defined by the POP quantification staging system receiving TVM or LSC mesh suspension were retrospectively recruited. Clinical evaluations before and 6 months after surgery included pelvic examination, urodynamic study, and a personal interview to evaluate urinary and sexual symptoms using questionnaires.

DETAILED DESCRIPTION:
All women with mainly uterine prolapse stage II or greater as defined by the POP-Q staging system receiving TVM or LSC mesh suspension surgeries at a tertiary referral center in Taiwan were included. The investigators excluded women with a hypertrophic uterus, huge fibroids, history of cervical dysplasia or endometrial pathology, history of postmenopausal bleeding in the past 12 months, and those unwilling to preserve their uterus. Concomitant mid-urethral sling operations were performed in women with current urodynamic stress incontinence unless the participants did not prefer a concomitant surgery. Cervical amputation was performed if the corpus/cervix ratio was less than 1 on the ultrasound. Concomitant anterior and posterior colporrhaphy were performed as needs.

The clinical evaluations consisted of a detailed history before and 6 months after surgery, including urinary analysis, pelvic examination using POP-Q system, urodynamic studies (UDS), transabdominal ultrasound, and personal interview to identify urinary and sexual symptoms with the Overactive Bladder Symptom Score (OABSS), the short forms of Urogenital Distress Inventory (UDI-6), the Incontinence Impact Questionnaire (IIQ-7), the Female Sexual Function Index (FSFI) questionnaire, and the Pelvic Organ Prolapse Distress Inventory (POPDI-6). Urinary symptoms with the standardized questionnaire taking into account the 2002 ICS definitions. The participants were asked to fill out the visual analog scale (VAS) scores during the postoperative day 1 round. Urodynamic studies, including non-instrumented uroflowmetry, filling and voiding cystometry, and urethral pressure profilometry, were performed according to the recommendations by the International Continence Society with a 6-channel urodynamic monitor (MMS; UD2000, Enschede, Netherlands). Any uninhibited detrusor contraction during filling cystometry was deemed positive for detrusor overactivity (DO).

As a follow-up, postoperative outpatient visits were at 1, 2, 3, 6, and 12 months and then semiannually beyond one year. Pelvic examination was performed routinely in every visit to clinics. Recurrence was defined as the most dependent portion of POP stage II or greater. The Clavien-Dindo grading was used for the classification of the intraoperative and postoperative complications of Long mesh surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with mainly uterine prolapse stage II or greater as defined by the POP-Q staging system

Exclusion Criteria:

* A hypertrophic uterus, huge fibroids
* History of cervical dysplasia or endometrial pathology
* History of postmenopausal bleeding in the past 12 months
* Unwilling to preserve their uterus

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with mainly uterine prolapse stage II or greater as defined by the POP-Q staging system
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | 12 months
  The POP-Q stage measurement after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yu Long, PhD, Principal Investigator — Kaohsiung Municipal University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016 Apr;27(4):655-84. doi: 10.1007/s00192-016-3003-y. PMID 26984443
- [Background] Korbly NB, Kassis NC, Good MM, Richardson ML, Book NM, Yip S, Saguan D, Gross C, Evans J, Lopes VV, Harvie HS, Sung VW. Patient preferences for uterine preservation and hysterectomy in women with pelvic organ prolapse. Am J Obstet Gynecol. 2013 Nov;209(5):470.e1-6. doi: 10.1016/j.ajog.2013.08.003. Epub 2013 Aug 3. PMID 23921090
- [Background] Wu MP, Long CY, Huang KH, Chu CC, Liang CC, Tang CH. Changing trends of surgical approaches for uterine prolapse: an 11-year population-based nationwide descriptive study. Int Urogynecol J. 2012 Jul;23(7):865-72. doi: 10.1007/s00192-011-1647-1. Epub 2012 Jan 24. PMID 22270728
- [Background] Long CY, Wang CL, Ker CR, Juan YS, Tsai EM, Lin KL. Laparoscopic Organopexy with Non-mesh Genital (LONG) Suspension: A Novel Uterine Preservation Procedure for the Treatment of Apical Prolapse. Sci Rep. 2018 Mar 20;8(1):4872. doi: 10.1038/s41598-018-23285-7. PMID 29559709
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2016 Oct 1;10(10):CD012376. doi: 10.1002/14651858.CD012376. PMID 27696355
- [Background] Long CY, Hsu CS, Wu CH, Liu CM, Wang CL, Tsai EM. Three-year outcome of transvaginal mesh repair for the treatment of pelvic organ prolapse. Eur J Obstet Gynecol Reprod Biol. 2012 Mar;161(1):105-8. doi: 10.1016/j.ejogrb.2011.12.007. Epub 2012 Jan 9. PMID 22226537
- [Background] Ker CR, Lin KL, Loo ZX, Juan YS, Long CY. Comparison of UpholdTM Vaginal Mesh Procedure with Hysterectomy or Uterine Preservation for the Treatment of Pelvic Organ Prolapse. Sci Rep. 2018 Jun 21;8(1):9438. doi: 10.1038/s41598-018-27765-8. PMID 29930249
- See also: U.S. Food and Drug Administration. Urogynecologic surgical mesh implants. — http://www.fda.gov/medical-devices/implants-and-prosthetics/urogynecologic-surgical-mesh-implants